CLINICAL TRIAL: NCT03390556
Title: Promoting Partnership and Improving Self-Management for Children With Persistent Asthma: A Pilot Program of Clinic-Based Asthma Education and Medication Labeling
Brief Title: Promoting Partnership and Improving Self-Management for Children With Persistent Asthma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rochester (Other)
Collaborators: New York State Department of Health (Other Government)
Responsible Party: Principal Investigator, Sean Frey, Assistant Professor, University of Rochester
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: RSRB00070365
Record Dates: First submitted 2017-12-15; First posted 2018-01-04 (Actual); Last update posted 2019-07-23 (Actual); Status verified 2019-07

CONDITIONS: Asthma in Children

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Asthma education (Experimental)
  Interventions: Other: Nurse-delivered education

INTERVENTIONS:
Other: Nurse-delivered education — The nurse will:
  1. Give the caregiver and child an overview of asthma, and discuss asthma control, triggers, and medications.
  2. Give caregivers information about asthma management written at or below 6th grade reading levels.
  3. Provide colored medication labels to distinguish controller from rescue medications following the action plan color scheme (green for controller medications, red for rescue medications). Teach-back methods will be used to elicit understanding of correct indications of use.
  4. Demonstrate MDI/spacer technique with teach-back.
  5. Discuss age-appropriate caregiver and child responsibility for asthma management within the family, with an overview of transitioning responsibility.
  6. Ask patients to make a 1 month follow-up appointment for asthma care.

SUMMARY:
The goal of this study is to evaluate a pilot of clinic-based intervention of asthma education. After a scheduled outpatient encounter for well-child care or asthma care has concluded, a pediatric nurse will teach participants (children and their caregivers) about asthma, provide clearly written information about how to manage asthma, and discuss how to manage asthma at home with cooperation between caregivers and children. Families will also receive current asthma prescriptions in clinic, and colored labels will be attached to medications in order to match the color scheme of asthma action plans (green labels for controller medications, red labels for rescue medications). Families will be followed for 3 months after the first clinic visit, including a follow-up visit in clinic 1 month later and a follow-up telephone call 3 months after starting. The nurse will reinforce key educational points and review medication use at the follow-up clinic visit. Families will also be invited to complete an additional in-depth interview following the 1 month clinic follow-up. The investigator hypothesizes that knowledge, self-efficacy, and reported adherence with asthma medications will increase for both caregivers and children/adolescents following the intervention and labeling of delivered medications. In addition, the investigator hypothesizes that children/adolescents will have more symptom free days and improved control following the intervention.

DETAILED DESCRIPTION:
Study Design:

The investigators propose a clinic-based intervention of asthma education and medication labeling to promote medication knowledge and self-efficacy for adherence among both caregivers and children. Approximately 40 children with uncontrolled persistent asthma and their caregivers will be enrolled prior to outpatient visits for asthma care (well child care or asthma-specific visits; total of 80 participants). After the scheduled encounter with a provider has concluded, enrolled dyads will receive an intervention of nurse-delivered asthma education and medication labeling. Dyads will then be followed prospectively for 3 months after the index visit. This follow-up period will include a clinic-based follow-up with a repeat of the intervention (1 month after enrollment, consistent with the follow-up interval suggested by national guidelines for uncontrolled asthma) and a second follow-up by telephone (2 months after clinic follow-up). Families will be invited to complete an additional in-depth interview following the 1 month clinic follow-up.

Subjects and Setting:

Children and adolescents 7-14 years of age will be screened for eligibility at a single ambulatory care location: the Golisano Children's Hospital Pediatric Practice, a National Committee for Quality Assurance (NCQA) accredited patient centered medical home (PCMH) in urban Rochester, New York. The investigators plan to enroll a convenience sample of 40 dyads of caregivers/children (total of 80 subjects) over an 8 month period. Children and adolescents will be enrolled equally from two age-based categories (7-10 years, 11-14 years). The range of child/adolescent ages is intended to select families with a range of shared responsibility for asthma medication use between the caregiver and child/adolescent. Some children independently use medications as early as six years old. On average, children bear half of the responsibility for controller medication use by age 11 years and have more responsibility than caregivers after age 13 years. Given these data, the specified age-based sub-groups are structured to reflect family dynamics in which children have <50% of responsibility for medications (7-10 years old) and ≥50% of responsibility for medications (11-14 years).

Study Procedures:

Screening Procedures: Screening will occur in a rolling fashion from January 2018 through August 2018. The investigators will identify potentially eligible children through a weekly review of pediatric clinic patients ages 7-14 years old who are (1) scheduled for well-child or asthma care over the following week, (2) have persistent asthma on their problem list, (3) have a current (within the last year) prescription for an inhaled controller medication, and (4) are covered by Medication or a Medicaid managed care program. After the reports are furnished, Dr. Frey will conduct a brief review of the patient's chart to determine whether key eligibility criteria are met (no known language barriers, no other significant medical or developmental conditions). Remaining eligibility criteria (i.e. determination of persistent/uncontrolled asthma per NHLBI guidelines) will be assessed during a single screening phone call prior to the scheduled visit, or by approaching caregivers at the time of scheduled visits if we are unable to reach caregivers by phone.

Baseline Assessment: The baseline survey assessment will be conducted following enrollment by the team research assistant within a private space in the clinic. All survey instruments will be available in English, and questions will be read aloud to the caregiver and child. If the baseline semi-structured survey is not completed before the provider encounter, caregivers will be given the option to complete the baseline either (a) before leaving clinic, or (b) over the telephone; completion in the clinic will be preferred so that children/adolescents can be separately interviewed in the presence of their caregivers.

Medication Selection and Delivery: Providers will be notified that their patients are enrolled into the program, and will be tasked with determining whether any changes in daily controller medications are indicated. The provider will electronically transmit prescriptions for both rescue and controller medications to the Strong Outpatient Pharmacy, located within the same building as the Pediatric Practice. All asthma prescriptions will be filled at this pharmacy during the trial in order to ensure that medications will be available for labeling in clinic, and parents will be informed of this during the consent process. The research assistant will call the pharmacy to notify them of new prescriptions; once these asthma prescriptions are filled, they pharmacy will send them to the Pediatrics Practice via the institution's pneumatic tube system. Any prescription medications that are not directly related to asthma management (including adjuvant therapies for allergic rhinitis) would be sent to the pharmacy of their choosing for normal processing and patient pick-up.

Nurse-delivered Education: The nurse will give the educational intervention after the provider encounter concludes. Nurses will be trained in intervention delivery and national asthma guidelines by Dr. Frey and Cindy Trubisky, Senior Director of Health Education for the American Lung Association (ALA) in Rochester, NY. This intervention will be directed toward both the caregiver and the child.

1. The nurse will give the parent and child a brief, scripted overview of asthma, and discuss asthma control, asthma triggers, and indications for using inhaled controller vs. rescue medications.
2. Parents will be given simple, written information about asthma and asthma management designed for low health-literacy audiences, specifically written at or below 6th grade reading levels, including:

   1. Information on appropriate metered dose inhaler (MDI)/ spacer technique
   2. An updated asthma action plan, with clear indications for when to use each inhaled medication (i.e., controller vs. rescue medications).
   3. A list of other local asthma resources and smoking cessation resources (as appropriate) will be given to caregivers
3. The nurse will provide colored medication labels to distinguish controller from rescue medications, following the action plan color scheme (green labels for controller medications, red labels for rescue medications). These labels will be applied to medications by the child/adolescent in clinic under nurse supervision.

   1. If medications are not filled in the Strong Outpatient Pharmacy and thus not available during the educational session, labels and instructions will be provided for patients to label medications at home. Care coordinators will follow-up with families to ensure appropriate labeling in this situation.
   2. Teach-back methods will be used to elicit understanding of correct indications of use for each medication (patient and caregiver).
4. The nurse will demonstrate the technique for MDI medications using a spacer, with teach-back performed by both the patient and caregiver.
5. They will discuss age-appropriate caregiver and child responsibility for asthma management within the family, with an overview of transitioning responsibility designed to reinforce the cooperative participation of both patients and caregivers.
6. Patients will be asked to make a 1 month follow-up appointment for asthma care.

Care Coordination: Pediatric practice care coordinators will contact all enrolled patient families by telephone 1 week prior to the scheduled follow-up appointment. In addition to functioning as a personalized reminder of the upcoming appointment, this phone call will also allow care coordinators to identify any surmountable barriers to scheduled care and remind families to bring all of the child's asthma medications to the visit.

Follow-Up Assessments: The study, including all follow-up assessments, will continue until the end of the 2018 calendar year. After the baseline assessment, each patient will have two additional follow-ups. The first will be completed in clinic, approximately 1 month (~4-6 weeks) after the baseline visit. As all enrolled patients will have symptomatic or poorly controlled persistent asthma, this follow-up interval is appropriate and supported by NHLBI guidelines.(2) A brief follow-up survey will be conducted prior to the provider encounter, and will include a repeat assessment of key measures from the baseline assessment. Additional asthma education will be repeated at this clinic visit, with a specific emphasis on reinforcing both the medication teaching and the importance of dyadic co-management. Asthma medication refills will be delivered to clinic and labeled with stickers as necessary. The second follow-up will occur approximately 2 months after the follow-up clinic visit (3 months after baseline), and will be a semi-structured interview conducted over the phone by the research assistant.

In-depth Interviews: During the clinic follow-up, caregivers and children will be invited to separately participate in in-depth interviews before leaving clinic; this use of qualitative research methods will allow for an enhanced understanding of family behaviors around medication management. The interview guide will specifically explore respondent thoughts on medication identification, the parent-to-child transfer of responsibility for medication use, and the usefulness of different intervention components. Interviews will be conducted in clinic if possible or over the phone if necessary; audio recordings will be transcribed. Thematic analysis will be conducted on interview transcripts until theoretical saturation is achieved within each subgroup of child/adolescent ages.

Compensation: Each participating caregiver/child dyad will receive $25 after completion of the initial baseline assessment and clinic visit in the form of a prepaid debit card. Participants will be paid an additional $25 after each follow-up assessment (one in clinic, one by phone), and a final payment of $25 will be available for any dyads that decide to participate in optional qualitative data collection (in-depth interviews). After the telephone follow-up, payment will be sent via mail. Total payment will be no more than $100 per dyad.

ELIGIBILITY:
Inclusion Criteria: (all 5 criteria must be met)

1. Physician diagnosis of asthma, based on review of medical records.
2. Uncontrolled asthma consistent with National Heart, Lung, and Blood Institute (NHLBI) guidelines, with at least 1 of the following based on caregiver report:

   a. If the child is 7-11 years old: i. An average of >2 days per week with asthma symptoms ii. >2 days per week with rescue medication use iii. >2 days per month with nighttime symptoms iv. ≥2 episodes of asthma during the past year that have required systemic corticosteroids b. If the child is 12-14 years old: i. An average of >2 days per week with asthma symptoms ii. >2 days per week with rescue medication use iii. Nighttime symptoms 1-3 times per week iv. ≥2 episodes of asthma during the past year that have required systemic
3. The child must have a current prescription (within the past year) of an inhaled asthma controller medication, such as an inhaled corticosteroid (ICS), based on review of electronic medical records.
4. The child/adolescent is between ≥7 and ≤14 years old.
5. The child/adolescent is insured by Medicaid or Medicaid managed care program.

Exclusion Criteria:

1. An inability to speak and understand English. Parents and children with low literacy / health-literacy skills will be eligible, as survey instruments will be administered verbally and educational materials will be designed for low-literacy populations.
2. No access to a working phone for follow-up, including care coordinator calls and the final follow-up survey.
3. Another significant medical condition identified in the child's medical record that could interfere with assessment of asthma control, including Cystic Fibrosis, congenital heart disease, or other chronic pulmonary disease.
4. A diagnosed developmental condition (e.g. Autism spectrum disorder or significant developmental delay) identified in the child's medical record that could impact the transition of responsibility for inhaled asthma medications from caregiver to child.
5. If the child or family is currently enrolled in a study conducted by The Preventive Care Program for Urban Children with Asthma (led by Dr. Jill Halterman).

Ages: 7 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 44 (Actual)
Dates: Start 2018-06-07 (Actual); Primary Completion 2019-05-31 (Actual); Study Completion 2019-06-30 (Actual)

PRIMARY OUTCOMES:
Change in caregiver self-efficacy from baseline to 1 month and 3 month follow-up | Baseline, 1 month follow-up, 3 month follow-up
  Parent asthma self-efficacy scale. This is a 13 item survey tool with 2 subscales: attack prevention (questions 1-6) and attack management (questions 7-13). For each question about perceived ability to manage asthma, parents select responses from a 5 point Likert scale (with 1 representing 'not at all sure' and 5 representing 'completely sure'). Responses to items in each subscale are averaged together to generate a subscale score. Higher mean subscale scores indicated increasing parent ability to perform asthma management tasks.
Change in child self-efficacy from baseline to 1 month and 3 month follow-up | Baseline, 1 month follow-up, 3 month follow-up
  Child asthma self-efficacy scale. This is a 14 item survey tool with 2 subscales: attack prevention (questions 1-8) and attack management (questions 9-14). For each question about perceived ability to manage asthma, children select responses from a 5 point Likert scale (with 1 representing 'not at all sure' and 5 representing 'completely sure'). Responses to items in each subscale are averaged together to generate a subscale score. Higher mean subscale scores indicated increasing child ability to perform asthma management tasks.
Change in caregiver reported adherence from baseline to 1 month and 3 month follow-up | Baseline, 1 month follow-up, 3 month follow-up
  Caregiver interview about adherence with controller medication over the previous 2 weeks. We will ask about the number of controller medication doses missed over the previous 2 weeks. As many children are instructed to use controller medications twice every day (once in the morning and once at night), the number of missed doses of controller medication ranges from 0 to 28 doses.
Change in child reported adherence from baseline to 1 month and 3 month follow-up | Baseline, 1 month follow-up, 3 month follow-up
  Child interview about adherence with controller medication over the previous 2 weeks. We will ask about the number of controller medication doses missed over the previous 2 weeks. As many children are instructed to use controller medications twice every day (once in the morning and once at night), the number of missed doses of controller medication ranges from 0 to 28 doses.

SECONDARY OUTCOMES:
Changes in caregiver report of symptom free days from baseline to 1 month and 3 month follow-up | Baseline, 1 month follow-up, 3 month follow-up
  We will ask how many full days (24 hours periods) that the patient was free of any asthma symptoms in the previous 2 weeks (range: 0-24 full days). A higher score indicates more days without symptoms.
Changes in child report of symptom free days from baseline to 1 month and 3 month follow-up | Baseline, 1 month follow-up, 3 month follow-up
  We will ask how many full days (24 hours periods) that the patient was free of any asthma symptoms in the previous 2 weeks (range: 0-24 full days). A higher score indicates more days without symptoms.
Changes in caregiver assessment of asthma control from baseline to 1 month and 3 month follow-up (children 12 years and older). | Baseline, 1 month follow-up, 3 month follow-up
  The asthma control test (ACT) is a validated asthma assessment tool for children and teens 12 years and older. This survey contains 5 questions, and assesses asthma symptoms over the previous 4 weeks. Answers range from 0 (indicating significant symptoms) to 5 (indicating no symptoms). The scale is interpreted through a sum score (range: 0-25 points), with a score of 20 points or higher indicating asthma control.
Changes in child assessment of asthma control from baseline to 1 month and 3 month follow-up (children 12 years and older). | Baseline, 1 month follow-up, 3 month follow-up
  The asthma control test (ACT) is a validated asthma assessment tool for children and teens 12 years and older. This survey contains 5 questions, and assesses asthma symptoms over the previous 4 weeks. Answers range from 0 (indicating significant symptoms) to 5 (indicating no symptoms). The scale is interpreted through a sum score (range: 0-25 points), with a score of 20 points or higher indicating asthma control.
Changes in caregiver and child asthma control from baseline to 1 month and 3 month follow-up (children ages 7-11 years) | Baseline, 1 month follow-up, 3 month follow-up
  The childhood asthma control test (cACT) is a validated asthma assessment tool for children 4 to 11 years old. This survey contains 7 questions, and assesses asthma symptoms over the previous 4 weeks. The first 4 questions about recent asthma symptoms are answered by children, with answers ranging from 0 (indicating significant symptoms) to 3 (indicating no symptoms). The final 3 questions are answered by parents, with answers ranging from 0 (indicating significant symptoms) to 5 (indicating no symptoms). The scale is interpreted through a sum score (range: 0-27 points), with a score of 20 points or higher indicating asthma control.

CONTACTS AND LOCATIONS:
Overall Officials: Sean M Frey, MD, MPH, Principal Investigator — University of Rochester
Locations (1):
- University of Rochester Medical Center, Rochester, New York, United States

IPD SHARING:
Plan to Share IPD: No